CLINICAL TRIAL: NCT00906087
Title: The Effect of Myocilin Genetic Variants on Intraocular Pressure and Blood Pressure Variation in Sitting and Supine Positions.
Brief Title: Effect of Myocilin Genetic Variants on Intraocular Pressure and Pressure Variation in Sitting and Supine Positions
Acronym: Myoc Gene
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sayoko E. Moroi, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Merck IISP#31911; Merck IISP#31911 (Other Grant/Funding Number: Merck)
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Glaucoma
Keywords: Myocilin gene; Glaucoma; dorzolamide and timolol combination eyedrop
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide-timolol combination; Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cosopt (Other): Intraocular pressure and blood pressure measurements will be compared under the following conditions: 1) after washout of clinical treatment, 2) after treatment with Cosopt, and 3) after another washout of Cosopt.
  Interventions: Drug: Cosopt (combination eyedrop of dorzolamide and timolol)

INTERVENTIONS:
Drug: Cosopt (combination eyedrop of dorzolamide and timolol) — One drop in each eye every twelve hours for six weeks
  Other Names: Cosopt

SUMMARY:
The purpose of this study is to determine if one of the genes that can cause glaucoma, called myocilin, are associated with larger eye pressure and blood pressure changes in sitting and lying down positions without glaucoma drug treatment and with glaucoma drug treatment with a combination medication called Cosopt® (Merck & Co., Inc.).

DETAILED DESCRIPTION:
Glaucoma is an important public health issue, and identifying new markers to improve treatment outcomes is a high priority. Progress in Mendelian genetic approaches has led to identifying 15 genes and 31 loci (http://www.ncbi.nlm.nih.gov/); however, since these monogenic forms of glaucoma are uncommon, other approaches are needed to identify genetic markers that contribute to common risk factors, such as elevated eye pressure, eye pressure fluctuation, and drug response variation.

It is well known that eye pressure varies over a 24-hour period,1-6 but the mechanisms that regulate this eye pressure rhythm are not yet fully known. Drance reported that 84% of normal eyes (N=320 eyes) had eye pressure fluctuations of less than 5 mmHg in contrast to only 6% of untreated glaucomatous eyes (N=138).7 Drance clearly recognized that eye pressure factors were more variable in eyes with glaucoma. Attention to this eye pressure fluctuation during glaucoma treatment is important because fluctuation leads to progression. The variation in eye pressure drug response profiles measured at selected times over a 24-hour period is related to the mechanism of action of these drugs, endogenous circadian rhythms, and glaucoma. The molecular and genetic tools are now available to identify potential genetic markers for these variable traits.

Advancing clinical research to the "translational" level is an important step to integrate our ever increasing knowledge base in genomics and proteinomics with clinical trials and clinical studies. Given the infrastructure at the University of Michigan with the strength in both glaucoma genetics and our resources in the clinic, it is possible to test for relationships between glaucoma genes and eye pressure. Although it is known that myocilin (MYOC) mutations cause the phenotype of high pressure open-angle glaucoma, the effect of these MYOC mutations in "pre-symptomatic" subjects and patients with early open-angle glaucoma on eye pressure variation is not known.

ELIGIBILITY:
Inclusion Criteria:

* Early OAG, as determined by a comprehensive ophthalmic examination
* Greater than or equal to 18 years of age
* Either gender
* Any race
* Both eyes meet eligibility criteria
* Cup to disc ratio less than 0.8 determined by fundoscopy and confirmed by disc photos
* Visual field parameters in the study eye: Pattern Standard Deviation (PSD) greater than 1.0 dB but less than 6.0 dB
* Ability to cooperate for an outpatient study involving at least five visits over a four month study period
* Ability to comply with Cosopt treatment regimen

Exclusion Criteria:

* Less than or equal to 18 years old
* Refusal to be genotyped or sign Informed Consent for Protocol 1991-144
* Pregnant or lactating women
* Medical conditions of severe pulmonary compromise with asthma or emphysema or cardiac contraindications to beta-blockers
* Ocular disease of chronic angle-closure glaucoma, iridocorneal endothelial disease, posterior polymorphous corneal dystrophy, epithelial downgrowth, uveitic glaucoma, or neovascular glaucoma
* Ocular surgery for glaucoma, including trabeculectomy, other glaucoma filtration surgery, glaucoma drainage implant, or laser cyclophotocoagulation
* Current use of systemic steroids or chemotherapeutic agents that non-selectively inhibit dividing cells
* Proliferative diabetic retinopathy, history of panretinal photocoagulation treatment, diabetic macular edema, or history of macular grid laser treatment
* History of changing treatment involving the use oral beta-blockers, angiotensin converting enzyme inhibitors, calcium channel blockers, or oral alpha 2-agonists in the prior two months or in the next month (i.e., must be on stable treatment with any of these drugs for at least two months)
* Patients taking erectile dysfunction drugs (i.e., Viagra, Cialis, Levitra)
* Contradictions:

  * bronchial asthma or a history of bronchial asthma
  * severe chronic obstructive pulmonary disease
  * sinus bradycardia
  * second or third degree atrioventricular block
  * overt cardiac failure
  * cardiogenic shock
  * hypersensitivity to any component of Cosopt

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-08-04 (Actual); Primary Completion 2012-07-18 (Actual); Study Completion 2012-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayoko E Moroi, MD, PhD, Principal Investigator — University of Michigan Department of Ophthalmology and Visual Sciences
Locations (1):
- W.K. Kellogg Eye Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cosopt: Cosopt 1 drop two times daily was administered for 6 weeks.
  Cosopt (combination eyedrop of dorzolamide and timolol): One drop in each eye every twelve hours for six weeks
Period: Initial Washout
Arm/Group | Cosopt
Started | 14
Completed Screening | 14
Begin Washout | 13
Completed Washout and Continue Protocol | 12
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1
Period: Cosopt Treatment 6 Weeks
Arm/Group | Cosopt
Started | 12
Completed | 12
Not Completed | 0
Period: Final Washout Period 4 Weeks
Arm/Group | Cosopt
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cosopt
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (19.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of males and females
  Participants
    Female | 4
    Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 14
Intraocular pressure right eye [Mean (Standard Deviation); unit: mmHg] — Baseline intraocular pressure = on current treatment
  mmHg
    Baseline at initial visit | 15.6 (2.10)
    After 4 week washout | 19.9 (4.33)
Intraocular pressure left eye [Mean (Standard Deviation); unit: mmHg]
  Baseline at initial visit | 16.4 (3.61)
  After 4 week washout | 20.4 (5.57)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure in Sitting and Supine Positions.
Description: Effect of Cosopt treatment on intraocular pressure changes in sitting to supine positions.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Cosopt: Intraocular pressure comparison after washout of Cosopt and while on treatment with Cosopt
  Cosopt (combination eyedrop of dorzolamide and timolol): One drop in each eye every twelve hours for six weeks
Arm/Group | Cosopt
Number analyzed (Participants) | 12
mmHg
  Sitting right eye | 18.5 (2.94)
  Sitting left eye | 19.4 (3.23)
  Supine right eye | 22.2 (3.06)
  Supine left eye | 22.8 (4.32)

2. Primary Outcome: Blood Pressure in Sitting to Supine Positions
Description: Effect of Cosopt treatment on blood pressure changes in sitting to supine positions.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Cosopt
Number analyzed (Participants) | 12
mmHg
  Sitting systolic blood pressure | 139.6 (20.40)
  Supine systolic blood pressure | 133.8 (21.7)
  Sitting diastolic blood pressure | 86.8 (12.29)
  Supine diastolic blood pressure | 89.3 (16.96)

3. Secondary Outcome: Myocilin Mutation Arg272Gly in Subjects
Description: Number of subjects with Myocilin Arg272Gly
Time Frame: 10 week study
Population: Only 1 participant had a MYOC mutation in the 3 exons
Measure: Count of Participants; unit: Participants
Arm/Group | Cosopt
Number analyzed (Participants) | 12
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 weeks of study participation (2 week washout; 6 weeks on Cosopt; 4 weeks washout)
Groups:
- Washout (no Glaucoma Medication): After appropriate washout, no glaucoma medication was administered for 6 weeks.
Arm/Group | Cosopt | Washout (no Glaucoma Medication)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cosopt (N=12) | Washout (no Glaucoma Medication) (N=14)
Eye pressure greater than 30 mmHg (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor wants an opportunity to review the data. I will send a PDF of this record on 3/17/2017.